CLINICAL TRIAL: NCT03608748
Title: Prospective Study: Early Detection of Advanced Fatty Liver Disease in the General Adult Population by Using Non-Alcoholic Fatty Liver Disease Score and Elastography
Brief Title: Early Detection of Advanced Fatty Liver Disease
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Rawi Hazzan, Head of Liver Unit, HaEmek Medical Center, Israel
Other Study IDs: 007-18-EMC
Record Dates: First submitted 2018-07-08; First posted 2018-08-01 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Non-alcoholic Fatty Liver Disease; Liver Fibrosis
Keywords: Nafld Score; Elastography
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Non-alcoholic fatty liver disease is the most common cause of chronic liver disease in the western world, affecting one in every three subjects.

The investigators hypothesize that a patient population without known liver disease has a certain percentage of patients with liver fibrosis who are undiagnosed and not monitored.

DETAILED DESCRIPTION:
The investigators will run an algorithm for the non-invasive diagnosis of advanced fibrosis in non-alcoholic fatty liver disease on a participants without known liver disease.

Nafld Score and Elastography are now being used to predict the severity of liver fibrosis and deciding whether the patient is going to a biopsy, clinical follow-up or further investigation of liver cirrhosis and complications.

The detection of participants with Nafld Score more than 0.675 (advanced fibrosis) will enroll them to an elastography test. Participants with advanced fibrosis according to elastography will be introduced to follow-up and treatment that should delay or prevent progression of the disease to more advanced conditions like: cirrhosis, portal hypertension, esophageal varicose veins and hepatocellular carcinoma.

If the investigators find that the results of the study are consistent with their hypothesis, this will lead to applying the flowchart to a larger sample of population in order to use it as a future survey.

Moreover, the investigators will check whether there is a correlation between Nafld Score and elastography in participants without know liver disease with Nafld Score more than 0.675.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 45-60 who belong to an initial clinic which was chosen arbitrarily.
2. Subjects without known liver disease.
3. Subjects agree to sign a consent form. -

Exclusion Criteria:

1. History of right-sided heart failure
2. History of liver disease including positive infectious serology for hepatitis B or C
3. Pregnant women
4. People incapable of judgment -

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All patients aged 45-60 years old without known liver disease who belong to an initial clinic which was chosen arbitrarily.
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Non-Alcoholic Fatty Liver Disease Score | Up to five minutes
  Non-alcoholic fatty liver disease Score (Nafld Score) is a non-invasive scoring system based on several laboratory tests that helps to estimate the amount of scarring in the liver. The score is made up of six parameters: age, BMI(body mass index), aspartate aminotransferase(AST) / alanine transaminase(ALT), platelet count, impaired fasting glucose(IFG), albumin.
  The Nafld Score formula is: -1.675 + 0.037 × age (years) + 0.094 × BMI (kg/m^2) + 1.13 × IFG/diabetes (yes = 1, no = 0) + 0.99 × AST/ALT ratio - 0.013 × platelets (×10^9/l) - 0.66 × albumin (g/dl).
  2 cutoff points were selected to identify the presence (> 0.675) and absence (< -1.455) of significant fibrosis.
  < -1.455: predictor of absence of significant fibrosis (F0-F2 fibrosis), negative predictive value 93% .
  between -1.455 and 0.675: indeterminate score.
  >0.675: predictor of presence of significant fibrosis (F3-F4 fibrosis), positive predictive value of 90%.
  The score will be calculated for all the participants.

SECONDARY OUTCOMES:
Elastography Test | Up to two hours
  Ultrasound Elastography is a non-invasive test which uses the technology of Shear Wave Elastography (SWE) obtained from the right liver lobe for staging liver fibrosis according to Metavir Fibrosis Score with sensitivity between 86% -98% and specificity between 90% -93%.
  Metavir Fibrosis Score is a system used to assess the extent of inflammation and fibrosis by histopathological evaluation in a liver biopsy.
  Liver fibrosis assessed by Shear Wave Elastography is well correlated to biopsy using Metavir Score.
  Participants with Nafld Score above 0.675 will undergo ShearWave Elastography.
  The outcome of the test will be correlated to Metavir Score system according to the chart below:
  SWE (kiloPascal) , METAVIR score, Fibrosis Level.
  Below 5 , F0 , No fibrosis.
  5.0-7.1 , F1 , Mild Fibrosis.
  7.1-8.7 , F2 , Significant Fibrosis.
  8.7-10.4 , F3 , Sever Fibrosis.
  10.4-19 , F4 , Cirrhosis.

CONTACTS AND LOCATIONS:
Overall Officials: Rawi Hazzan, Dr, Principal Investigator — haemek medical center
Locations (1):
- Haemek medical center, Afula, Israel